CLINICAL TRIAL: NCT04838171
Title: Investigation of White Blood Cells to Support the Development of Engineered Regulatory T Cell (Treg) Therapies
Brief Title: Prospective Study of White Blood Cells
Status: Recruiting | Type: Observational
Sponsor: Quell Therapeutics Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: QEL-RP-001
Record Dates: First submitted 2021-04-01; First posted 2021-04-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Autoimmune Diseases; Inflammation; Rejection; Transplant, Liver
MeSH Terms: conditions — Autoimmune Diseases; Inflammation; Rejection, Psychology | interventions — Leukocyte Count

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Specimen collection to support development of engineering Treg
  Interventions: Other: White blood cell and blood collection

INTERVENTIONS:
Other: White blood cell and blood collection — Mononucleocytes will be collected via apheresis

SUMMARY:
The purpose of this study is to investigate white blood cells from volunteering donors to support the development of engineered regulatory T cell therapies.

ELIGIBILITY:
No additional inclusion/ exclusion criteria will be applied by Quell other than those specified by the consenting institutions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Volunteers willing to provide white blood cells for research.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
WBC characterisation to support the development of engineered regulatory T cells. | 5 years
  number, type and function of white blood cells in healthy controls and in patients

CONTACTS AND LOCATIONS:
Locations (1):
- Quell Investigator Site 01, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No